CLINICAL TRIAL: NCT00888693
Title: A Multiple Dose Study of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ABT-288 in Stable Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Hana Florian, MD/Associate Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M10-752
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2010-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — 2-(4'-(5-methylhexahydropyrrolo(3,4-b)pyrrol-1-yl)biphenyl-4-yl)-2H-pyridazin-3-one

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- 1 (Experimental): ABT-288 vs placebo capsules administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 2 (Experimental): ABT-288 vs placebo capsules administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 3 (Experimental): ABT-288 vs placebo capsules administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 4 (Experimental): ABT288 vs placebo administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 5 (Experimental): ABT-288 vs placebo administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 6 (Experimental): ABT-288 vs placebo administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 7 (Experimental): ABT-288 vs placebo administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 8 (Experimental): ABT-288 vs placebo administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo
- 9 (Experimental): ABT-288 vs placebo administered orally once daily for 14 days
  Interventions: Drug: ABT-288; Drug: Placebo

INTERVENTIONS:
Drug: ABT-288 — See Arm Description for details.
Drug: Placebo — See Arm Description for details.

SUMMARY:
Evaluate the safety, tolerability and pharmacokinetics of ABT-288 in order to determine the maximum tolerated dose of ABT-288 in stable schizophrenic volunteers receiving treatment with an atypical antipsychotic.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed informed consent;
* Current DSM-IV-TR diagnosis of schizophrenia;
* Clinically stable on the same single second-generation antipsychotic for the past 8 weeks;
* Meets study-specific PANSS criteria;
* Willing and able to cooperate with cognitive testing
* Females are not pregnant, not breast-feeding;
* Females are post-menopausal or surgically sterile or practicing birth control;
* Males are surgically sterile or agree to be sexually inactive or use barrier method of birth control

Exclusion Criteria:

* Subject has a substance dependence disorder that has not been in sustained remission for at least 1 year;
* Diagnosis of schizoaffective disorder;
* Bipolar disorder, manic episode, dementia, OCD, or drug-induced psychosis or current major depressive disorder;
* Diagnoses with mental retardation; acute psychosis hospitalization within past 6 months;
* Current clozapine treatment; suicidal ideation or behavior;
* BMI of 39 or greater; current homicidal or violent ideation;
* Medical or CNS condition other than schizophrenia that could affect cognitive performance or testing; relevant drug sensitivity or allergy; positive urine screen for alcohol or drugs of abuse;
* Positive hepatitis or HIV test result;
* Recent clinically significant illness/infection or surgery;
* Recent blood product transfusion, donation or loss of 5 mL/kg of blood;
* Visual, hearing or communication disability

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Physical Exams, Brief Neurological Exams, Vitals, Orthostatic Vitals, ECG, Laboratory tests, | Days -1 to 21
Pharmacokinetics; optional CSF for arms 7, 8 & 9 | Days -1 to 21

SECONDARY OUTCOMES:
Extrapyramidal Symptom Rating Scale | Day -1, Day 14
Columbia Suicide Severity Rating Scale | Screening, Day 15
Pharmacodynamics: CANTAB & PANSS | Screening, Day -1, Day 14
Pharmacodynamics: Pittsburgh Sleep Quality Index-Modified | Day -1, Day 15

REFERENCES:
- [Background] Othman AA, Haig G, Florian H, Locke C, Gertsik L, Dutta S. The H3 antagonist ABT-288 is tolerated at significantly higher exposures in subjects with schizophrenia than in healthy volunteers. Br J Clin Pharmacol. 2014 Jun;77(6):965-74. doi: 10.1111/bcp.12281. PMID 24215171